CLINICAL TRIAL: NCT07102121
Title: Comparison of Post Cementation Sensitivity Between Resin-Modified Glass Ionomer Cement and Conventional Glass Ionomer Cement as a Luting Material: A Randomized Clinical Trial
Brief Title: Comparison of Post Cementation Sensitivity Between RMGIC and GIC as Luting Materials in a Randomized Clinical Trial
Acronym: RMGICvsGIC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saidu College of Dentistry (Other)
Responsible Party: Principal Investigator, Dr Ajmal Khan, saiduCDentistry, Saidu College of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8643/SCD/SWAT/ethical
Record Dates: First submitted 2025-07-25; First posted 2025-08-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Dental Pulp Disease; Dental Pain and Sensation Disorder
Keywords: sensitivity; cementation; post cementation
MeSH Terms: conditions — Dental Pulp Diseases; Toothache; Sensation Disorders; Hypersensitivity | interventions — Glass Ionomer Cements

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment intervention model, where participants are randomly allocated into two groups in a 1:1 ratio. One group will receive resin-modified glass ionomer cement (RMGIC) and the other will receive conventional glass ionomer cement (GIC) for luting fixed dental prostheses. Each participant will undergo a standardized clinical procedure including tooth preparation, isolation, and cementation by trained postgraduate trainees. The intervention (type of cement) is applied once, and post-cementation sensitivity will be assessed at 24 hours and 7 days following the procedure. Randomization and stratification will be employed to reduce bias and ensure comparability between groups
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, masking will be applied to the participants and the outcomes assessor to reduce performance and detection bias. Participants will not be informed about the type of luting cement used during their treatment. The outcomes assessor, responsible for evaluating post-cementation sensitivity, will also be blinded to group allocation to ensure unbiased data collection. However, due to the clinical differences in handling the materials, the care providers and investigators cannot be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Glass Ionomer Cement (RMGIC) (Active Comparator): Participants in this group will receive fixed prostheses cemented with resin-modified glass ionomer cement (RMGIC) according to manufacturer's instructions. Tooth preparation will be carried out by postgraduate trainees, and cementation will include light curing of RMGIC for 10 seconds using an LED light. Sensitivity will be assessed at 24 hours, one week, 1 month, 2 months and 3 months post-cementation
  Interventions: Procedure: luting material applaication with Modified Glass Ionomer Cement (RMGIC)
- Conventional Glass Ionomer Cement (GIC) (Active Comparator): Participants in this group will receive fixed prostheses cemented with conventional glass ionomer cement (GIC). Tooth preparation and cementation will be performed by the same protocol as the other arm, except no light curing will be involved. Sensitivity levels will be recorded at 24 hours, one week , one month, two months and three months after cementation.
  Interventions: Procedure: luting material applaication with Modified Glass Ionomer Cement (RMGIC)

INTERVENTIONS:
Procedure: luting material applaication with Modified Glass Ionomer Cement (RMGIC) — The intervention involves the use of two different types of luting cements-resin-modified glass ionomer cement (RMGIC) and conventional glass ionomer cement (GIC)-for the cementation of fixed dental prostheses. The objective is to compare post-cementation sensitivity between the two materials. All clinical procedures, including tooth preparation, isolation, and cementation, will follow standardized protocols. Sensitivity will be measured using the Visual Analog Scale (VAS) at 24 hours and 7 days post-procedure. The study will maintain consistency across both groups, with the only variable being the type of cement used.
  Other Names: luting material applaication with Glass Ionomer Cement GIC)

SUMMARY:
This randomized controlled trial aims to compare post-cementation sensitivity between resin-modified glass ionomer cement (RMGIC) and conventional glass ionomer cement (GIC) as luting materials. Conducted at the Prosthodontics Department, Saidu College of Dentistry, Swat, the study will enroll 248 patients aged 15-70 with vital abutment teeth, randomly assigned to receive either RMGIC or GIC. Sensitivity will be assessed using a 10-point Visual Analog Scale (VAS), with scores above 1 considered indicative of post-operative sensitivity and further categorized for analysis. Strict inclusion/exclusion criteria and randomization will control bias and confounders. Data will be analyzed in SPSS 22 using t-tests and chi-square tests, with significance set at p≤0.05.

DETAILED DESCRIPTION:
Dental prostheses are frequently used to replace missing teeth. Fixed partial dentures are regarded as the gold standard for restoring lost teeth, aiming to recover proper function, speech, and appearance. These fixed prostheses must be securely attached to the neighboring teeth using specific bonding agents known as luting cements. Ideal luting materials should exhibit low solubility, biocompatibility, resistance to leakage, and should not cause discomfort or sensitivity after cementation. Common luting agents include glass ionomer cement (GIC), resin-modified glass ionomer cement (RMGIC), zinc phosphate cement, and zinc oxide eugenol cement. Among these, GIC and RMGIC are considered reliable and long-lasting choices for luting purposes.

This randomized controlled trial aims to compare post-cementation sensitivity between resin-modified glass ionomer cement (RMGIC) and conventional glass ionomer cement (GIC) as luting materials. Conducted at the Prosthodontics Department, Saidu College of Dentistry, Swat, the study will enroll 248 patients aged 15-70 with vital abutment teeth, randomly assigned to receive either RMGIC or GIC. Sensitivity will be assessed using a 10-point Visual Analog Scale (VAS), with scores above 1 considered indicative of post-operative sensitivity and further categorized for analysis. Strict inclusion/exclusion criteria and randomization will control bias and confounders. Data will be analyzed in SPSS 22 using t-tests and chi-square tests, with significance set at p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 15 to 70 years

Both male and female participants

Abutment teeth with vital pulp

Sound abutment teeth with no signs of attrition, erosion, or abrasion

No history of pulp capping procedures on abutment teeth

Exclusion Criteria:

* Patients currently undergoing orthodontic treatment or who completed it within the last 3 months

Use of bleaching or desensitizing agents

History of recent periodontal surgery

Patients on medications that affect pain perception (e.g., analgesics, carbamazepine)

Patients with psychiatric conditions that may affect pain reporting or compliance

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 496 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
Dentinal sensitivity | At 24 hours, one week, one month, 2 months and three months after cementation
  Patient-reported sensitivity will be assessed using a 10-point Visual Analog Scale (VAS), where 0 indicates no pain/sensitivity and 10 indicates the worst possible pain/sensitivity. A VAS score greater than 1 will be considered as post-cementation sensitivity. The scores will also be categorized as:
  No sensitivity: VAS 0-1
  Mild: VAS 2-3
  Moderate: VAS 4-7
  Severe: VAS 8-10

CONTACTS AND LOCATIONS:
Locations (1):
- Dental college, Mingora, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
For ethical issue